CLINICAL TRIAL: NCT02940769
Title: Neurobiological Effects of Light on MDD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding no longer available
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Juan Francisco Lopez, Associate Professor Emeritus, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PRITZ1
Record Dates: First submitted 2015-09-22; First posted 2016-10-21 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Major Depressive Disorder
Keywords: depression; insomnia; light; cortisol; melatonin
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- light glasses (Experimental): Study subjects will wear light glasses
  Interventions: Device: light glasses
- sham glasses (placebo) (Sham Comparator): Study subjects will wear sham glasses
  Interventions: Device: sham glasses (placebo)

INTERVENTIONS:
Device: light glasses — light glasses
  Arms: light glasses
Device: sham glasses (placebo) — sham light glasses
  Arms: sham glasses (placebo)

SUMMARY:
The primary study objective is to observe/measure the circadian pattern of sleep, Cortisol and Melatonin in MDD subjects and Control subjects. We will also assess if controlled exposure to light in MDD subjects (post-partum females, non- post-partum females and males) will change these parameters using light glasses. In addition to the biological outcome measures (sleep, cortisol and melatonin) we will also monitor sleep and depressive symptoms in the research subjects for the duration of the protocol.

DETAILED DESCRIPTION:
In this study we will collect baseline hormone data and clinical data along with assessing light exposure using a Daysimeter in MDD participants and control subjects. We will collect baseline Daysimeter data for 5 days and then collect cortisol and melatonin levels in both MDD subjects and Control Subjects. Control subjects will complete the study following the sample collection. MDD participants will then have a light intervention (sham or active).

Following the Daysimeter and hormone data collection, MDD subjects in each group will be randomly assigned into a non-treatment group or treatment group. While continuing to wear the Daysimeter, all MDD subjects will wear assigned glasses for 2 hours prior to bedtime. The subject will choose the bedtime hour and try and consistently wear the glasses at the same time throughout the study. Subjects will then wear the assigned glasses in the am upon waking for 1 hour. Following 7 days wearing the assigned glasses MDD subjects will repeat the sample collection for Cortisol and Melatonin

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent before beginning any study-specific procedures
2. Male and female patients at least 18-60 years of age
3. Women with reproductive potential must have a negative pregnancy test;
4. Meets DSM-IV criteria for Major Depressive disorder
5. Hamilton Depression Rating Scale total score of 15 or greater
6. Negative Drug screen for drugs of abuse
7. No sleep altering medications, including herbal preparations. If subjects previously taking any of these medications, they need to be 1 week off of medications before starting the study.
8. If currently on SSRI, subjects must have been on them for 6-8 weeks.
9. PSQI of >5 and without sleep difficulties unrelated to the depression

Exclusion criteria:

MDD subjects will be excluded if:

1. Subjects with a comorbid current primary Axis I disorder of OCD, Eating disorder or any non-anxiety related Axis 1 diagnosis.
2. Subjects who meet DSM-IV criteria for substance dependence confirmed by the SCID, for any substance except nicotine, within 3 months of screening.
3. Subjects who meet DSM-IV criteria for substance abuse within 3 months of screening.
4. Subjects with positive urine toxicology screen for illicit substances of abuse (aside from cannabis, if patient not abusing and agrees to stop use).
5. Subjects with a history of clinically significant cardiac, renal, neurologic, cerebrovascular, metabolic, or pulmonary disease, or other disease or clinical findings that are unstable, or that in the opinion of the investigator, would confound biological assessments.
6. Female subjects who are pregnant or who are breastfeeding or planning to become pregnant during the study.
7. Subjects who, in investigator's opinion, would be non-compliant with the study procedures
8. Subjects with current psychotic symptoms (delusions or hallucinations).
9. Existing sleep problems unrelated to the depression
10. Potential study subjects who are actively suicidal

Healthy Volunteers must fulfill all of the following inclusion criteria:

1. Able to provide informed consent before beginning any study-specific procedures
2. Not meet a current or lifetime DSM-IV Axis I disorder

2) Male and female patients at least 18 years of age 3) Women with reproductive potential must have a negative pregnancy test; 4) Medication free, including herbal medications 5) Negative drug screen for drugs of abuse. 6) PSQI of < 5

Healthy volunteers will be excluded if:

1. A current or lifetime DSM-IV Axis I disorder.
2. A positive urine toxicology screen for illicit substances of abuse (aside from cannabis, if not abusing and agrees to stop use).
3. A history of clinically significant cardiac, renal, neurologic, cerebrovascular, metabolic, or pulmonary disease, or other disease or clinical finding that is unstable or that, in the opinion of the investigator, would confound biological assessments.
4. Females who are pregnant, breastfeeding or planning to become pregnant during the study.
5. People who, in investigator's opinion, would be non-compliant with the study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
salivary cortisol levels | Change is being assessed over time following the intervention (day 5, day 6, day 12 & day 13)

SECONDARY OUTCOMES:
salivary melatonin levels | Change is being assessed over time following the intervention (day 5, day 6, day 12 & day 13)

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Lopez, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No